CLINICAL TRIAL: NCT00841321
Title: Ginkgo Biloba for Cognitive Impairment in Multiple Sclerosis
Brief Title: Trial of Ginkgo as a Treatment for Cognitive Problems in Multiple Sclerosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: B4368-R
Record Dates: First submitted 2009-02-09; First posted 2009-02-11 (Estimated); Results first posted 2014-05-05 (Estimated); Last update posted 2014-06-06 (Estimated); Status verified 2014-05

CONDITIONS: Multiple Sclerosis; Cognitive Ability, General
Keywords: Ginkgo biloba; Multiple Sclerosis; Cognition; Neuropsychological Tests; Neurobehavioral Manifestations; Quality of life; Randomized Controlled Trials; Placebos; Double-Blind Method
MeSH Terms: conditions — Multiple Sclerosis; Neurobehavioral Manifestations | interventions — Ginkgo Extract; Ginkgo biloba extract

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm 1 (Active Comparator): Subjects with multiple sclerosis and documented cognitive impairment will be randomized to take the intervention or placebo.
  Interventions: Drug: Ginkgo biloba
- Arm 2 (Placebo Comparator): Subjects with multiple sclerosis and documented cognitive impairment will be randomized to receive the placebo.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ginkgo biloba — 120 mg orally twice a day for 12 weeks
  Other Names: EGb 761
  Arms: Arm 1
Drug: Placebo — One capsule orally twice a day for 12 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to see if treatment with Ginkgo improves cognitive function in people with multiple sclerosis who have cognitive problems.

DETAILED DESCRIPTION:
Objectives:

Primary objective: Determine the difference between subjects treated with Ginkgo biloba (GB) and subjects treated with placebo for 12 weeks on the performance of a battery of neuropsychological tests that are frequently impaired in Multiple Sclerosis (MS): the Stroop test, the Paced Auditory Serial Addition Test (PASAT), the California Verbal Learning Test (CVLT-II), and the Controlled Oral Word Association Test (COWAT). Secondary objectives: Determine the difference between the two groups after treatment in the following outcomes: 1) incidence of treatment related side effects, 2) cognitive performance as reported by the subjects on the Perceived Deficits Questionnaire, 3) cognitive performance as reported by the subject's family members or caregivers as measured on the Multiple Sclerosis Neuropsychological Screening Questionnaire and 4) community integration as measured with the Community Integration Questionnaire.

Research plan:

This will be a randomized double blind placebo controlled trial of GB 120 mg twice a day for 12 weeks.

Methods:

One hundred fifty-eight subjects (79 per group) will be randomly assigned to placebo or GB. Subjects will be evaluated at baseline and exit with the cognitive test battery and the self report measures detailed above.

For the primary outcome, multivariate analysis of covariance (MANCOVA) will be used to analyze the changes in all the cognitive tests simultaneously. This analysis will be followed by the analysis of covariance (ANCOVA) for each of the cognitive tests in the battery. The sample size we selected has a power of 0.80 with an alpha level of 0.05 on the overall MANCOVA and for each of the ANCOVA's after Bonferroni's correction.

The self report measures will be analyzed using ANCOVA with baseline responses as covariates.

Safety evaluations will include complete blood count and metabolic panel as well as physical exams at baseline and at exit. The physical exam will include the Expanded Disability Scale (EDSS). Telephone follow-ups will be done monthly while on treatment and one month after exiting the study to review study procedures and assess side effects. Adverse reactions will be classified using the categories and grading in the Cancer Therapy Evaluation Program (CTEP) Common Toxicity Criteria (CTC) Version 3.0 and reported to the Institutional Review Board (IRB) following the institutions guidelines. A Data Safety Management Board (DSMB) will oversee the study.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of multiple sclerosis by McDonald's criteria
* Age 18 to 65 years, inclusive
* A score minus one standard deviation below the mean on one or more of the following tests: PASAT, COWAT, CVLT-II, Stroop
* EDSS 0 - 7.5, inclusive
* No Ginkgo biloba in preceding 30 days
* Native English speaker

Exclusion Criteria:

* Current substance abuse disorder, psychosis, or significant depression (score on the Beck Depression Inventory II (BDI -II) greater than 28
* Any significant uncontrolled medical problem including diabetes requiring insulin
* Relapse of multiple sclerosis within the 30 days before screening
* Abnormalities of coagulation or current use of anticoagulants or antiplatelet agents
* Elective surgery planned for the study period or the following four weeks
* Epilepsy or history of seizures
* Use of nifedipine, nicardipine, Saint John's Wort, papaverine, mono amine oxidase inhibitors
* Pregnancy or women not using a reliable form of contraception
* Corrected binocular visual acuity worse than 20/50 or more than one error on binocular color vision testing with the Ishihara Color Plates or sustained nystagmus or diplopia on primary gaze
* Inability to complete the neuropsychological test battery at the screening visit
* History of alcohol abuse or illicit drug use in the prior six months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2009-01; Primary Completion 2010-11 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis N. Bourdette, MD, Principal Investigator — Portland VA Medical Center, Portland, OR
Locations (2):
- United States (2):
  - Portland VA Medical Center, Portland, OR, Portland, Oregon
  - VA Puget Sound Health Care System, Seattle, Seattle, Washington

REFERENCES:
- [Result] Lovera JF, Kim E, Heriza E, Fitzpatrick M, Hunziker J, Turner AP, Adams J, Stover T, Sangeorzan A, Sloan A, Howieson D, Wild K, Haselkorn J, Bourdette D. Ginkgo biloba does not improve cognitive function in MS: a randomized placebo-controlled trial. Neurology. 2012 Sep 18;79(12):1278-84. doi: 10.1212/WNL.0b013e31826aac60. Epub 2012 Sep 5. PMID 22955125
- [Derived] Hughes AJ, Parmenter BA, Haselkorn JK, Lovera JF, Bourdette D, Boudreau E, Cameron MH, Turner AP. Sleep and its associations with perceived and objective cognitive impairment in individuals with multiple sclerosis. J Sleep Res. 2017 Aug;26(4):428-435. doi: 10.1111/jsr.12490. Epub 2017 Jan 17. PMID 28093823
- See also: Department of Veteran Affairs MS Centers of Excellence — http://www.va.gov/ms/
- See also: MS Center of Oregon — http://www.ohsu.edu/xd/research/centers-institutes/neurology/multiple-sclerosis-center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study sites were the Portland VA Medical Center, Portland, Oregon & VA Puget Sound Health Care System, Seattle Washington. Enrollment time span was January 2009 to November 2010.
Pre-assignment Details: A total of 172 people were assessed for eligibility and 52 did not meet criteria for randomization. Reasons for exclusion included cognitive scores too high (35), Beck Depression Inventory II scores too high (7), failed color vision test(4), usage of contraindicated medications (2); miscellaneous reasons (4).
Groups:
- Placebo: Placebo, one capsule orally twice a day for 12 weeks.
- Ginkgo: Ginkgo (EGb-761), 120-mg tablet of ginkgo twice a day for 12 weeks.
Period: Overall Study
Arm/Group | Placebo | Ginkgo
Started | 59 | 61
Completed | 58 | 58
Not Completed | 1 | 3
Not completed — Lost to Follow-up | 1 | 1
Not completed — Adverse Event | 0 | 2

BASELINE CHARACTERISTICS:
Population: Based on pilot data (compliance of 80%,dropout rate of 20%) the estimated sample size needed to power the study was 158 enrolled to yield 110 with complete observations. In this study, enrollment was stopped at 121 participants with more than 110 subjects completing the study (dropout rate less than 5%).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Ginkgo | Total
Number analyzed (Participants) | 59 | 61 | 120
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 59 | 61 | 120
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.0 (9.5) | 51.3 (8.6) | 52.1 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 37 | 29 | 66
  Male | 22 | 32 | 54
Race/Ethnicity, Customized [Number; unit: participants]
  White | 59 | 55 | 114
  Non-white | 0 | 6 | 6
Disease duration, average number of years [Mean (Standard Deviation); unit: years] — For each group the average number of years that participants had Multiple Sclerosis
  years | 19.3 (11.8) | 20.9 (11.8) | 20.1 (11.8)
Expanded Disability Status Scale [Mean (Standard Deviation); unit: units on a scale] — 0:Normal
  1. No disability(dis) 1.5:(min)signs
  2. Min dis
  3. Moderate(mod) dis
  4. Amb no aid>=500 m 4.5:>=300 m
  5. >=200 m 5.5:>=100 m
  6. Amb unilateral aid>=100 m 6.5:Amb bilateral aid>=20 m
  7. Amb < 5 m 7.5:Unable to take few steps
  8. Bedbound, uses of arms 8.5:Bedbound some use of arms & some self care
  9. Helpless in bed 9.5:Unable to communicate/eat/swallow
  10. Dead
  units on a scale | 4 (2) | 4 (2) | 4 (2)
Type of Multiple Sclerosis [Number; unit: Participants]
  Primary Progressive MS | 4 | 5 | 9
  Progressive Remitting MS | 1 | 0 | 1
  Relapsing Remitting MS | 35 | 42 | 77
  Secondary Progressive MS | 19 | 14 | 33

OUTCOME MEASURES:

1. Primary Outcome: Primary Outcome is Performance on the Interference Condition of the Stroop, the Long Delay Free Recall Portion of the California Verbal Learning Test II, the 2 Second Paced Auditory Serial Addition Test and the Controlled Oral Word Association Test.
Description: Performance at exit adjusted for baseline performance on 4 neuropsychological tests:
  STROOP(Victoria version):Tests attention&executive function. Outcome is the interference condition condition; time needed to name the colors in which words (which are names of colors) are printed. Words and colors are mismatched.
  CaliforniaVerbalLearningTest- II: Tests verbal/learning/memory. Outcome number of words (shopping list) remembered after 20 min delay with no cues.
  PacedAuditorySerialAdditionTest:Tests working memory/sustained attention. Outcome is the number of correct responses to recording giving numbers every 2 sec. Last 2 numbers must be added together before the next number.
  ControlledOralWordAssociationTest:Tests letter fluency. Outcome number of words produced in one minute for each of 3 letters.
  Measures reported as Z-scores based on the available population norms for each test; range -infinite +infinite; 0 average; -1=1std below average; +1=1std above average.
Time Frame: 12 weeks
Population: Data of all 120 participants was analyzed. For subjects with missing exit values (1 placebo, 2 ginkgo) the baseline measures were carried forward in the analysis.
Measure: Mean (Standard Deviation); unit: z-scores
Groups:
- Ginkgo Baseline; Ginkgo Exit: Ginkgo (EGb-761), 120-mg tablet of ginkgo twice a day for 12 weeks.
- Placebo Baseline; Placebo Exit: Placebo, one capsule orally twice a day for 12 weeks.
Arm/Group | Ginkgo Baseline | Ginkgo Exit | Placebo Baseline | Placebo Exit
Number analyzed (Participants) | 61 | 61 | 59 | 59
z-scores
  PASAT | -1.4 (0.8) | -1.3 (0.9) | -1.2 (0.9) | -1.0 (1.1)
  Stroop Interference | -0.9 (1.6) | -0.8 (1.8) | 01.0 (1.4) | -0.3 (1.1)
  COWAT | -0.9 (1.0) | -0.7 (1.0) | -1.0 (1.0) | -0.8 (1.0)
  CVLT-II delayed free recall | -0.5 (1.2) | -0.4 (1.2) | -0.5 (1.2) | -0.4 (1.2)
Statistical Analysis 1: Comparison: Ginkgo Exit vs Placebo Exit; PASAT Exit Z-score least square means difference adjusted for baseline. Positive values indicate a beneficial effect from treatment with Ginkgo; Test type: Superiority or Other; p = .1, ANCOVA — Nominal value. Per protocol univariate tests would only be considered significant in the multivariate test was significant; Mean Difference (Final Values) = -0.2, 95% CI 2-sided [-0.5 to 0.1], Standard Error of Mean 0.15
Statistical Analysis 2: Comparison: Ginkgo Exit vs Placebo Exit; Stroop Exit Z-score least square means difference adjusted for baseline.Positive values indicate a beneficial effect from treatment with Ginkgo; Test type: Superiority or Other; p = 0.007, ANCOVA — Not adjusted for multiple comparison. Nominal value. Per protocol univariate tests would only be considered significant in the multivariate test was significant; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Ginkgo Exit vs Placebo Exit; COWAT Exit Z-score least square means difference adjusted for baseline. Positive values indicate a beneficial effect from treatment with Ginkgo; Test type: Superiority or Other; p = 0.5, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.2 to 0.3], Standard Error of Mean 0.1
Statistical Analysis 4: Comparison: Ginkgo Exit vs Placebo Exit; CVLT-II Delayed Recall Exit Z-score least square means difference adjusted for baseline. Positive values indicate a beneficial effect from treatment with Ginkgo; Test type: Superiority or Other; p = 0.5, ANCOVA — [p-value comment as in outcome 1, analysis 2]; Mean Difference (Final Values) = 0, 95% CI [-0.3 to 0.3], Standard Error of Mean 0.15
Statistical Analysis 5: Comparison: Ginkgo Exit vs Placebo Exit; MANCOVA for all four cognitive tests at exit adjusting for baseline. Individual ANOVAs were to follow if the multivariate test was significant; Test type: Superiority or Other; p = 0.19, MANCOVA; MANCOVA

2. Secondary Outcome: Secondary Outcome: Measures of Self-report as Well as Family Reports of Subject's Cognitive Deficits and Assessment of Social Integration.
Description: The Perceived Deficits Questionnaire (PDQ), a standardized questionnaire in which the subject reports on his or her cognitive function; Measure total score Range (0 best - 80 worse) Multiple Sclerosis Neuropsychological Screening Questionnaire (MSNQ), in which the family member who was most aware of the participant's cognitive deficits reports on the subject's cognitive deficits; measure total score range (0 best - 60 worse) 'and the Community Integration Questionnaire (CIQ) in which the subject reports his or her degree of social integration; range (0 worst - 32 best); measure total score.
  Sub-scales for these 3 measures were not used for outcome measures only total scores.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Ginkgo Baseline | Ginkgo Exit | Placebo Baseline | Placebo Exit
Number analyzed (Participants) | 61 | 61 | 59 | 59
units on a scale
  PDQ: Perceived deficits Questionnaire | 37.2 (11.5) | 31.7 (11.1) | 38.2 (13.8) | 33.4 (15.7)
  MSNQ: MS Neuropsychological ScreeningQuestionnaire | 25.2 (11.1) | 24.5 (11.1) | 27.8 (12.5) | 27.0 (11.1)
  CIQ:Community Integration Questionnaire | 23.0 (3.7) | 23.1 (4.4) | 23.0 (4.5) | 22.9 (4.4)
Statistical Analysis 1: Comparison: Ginkgo Exit; Perceived Deficits Questionnaire; Test type: Superiority or Other; p = 0.4, ANCOVA; Mean Difference (Final Values) = -0.5, 95% CI 2-sided [-5.7 to 4.7], Standard Error of Mean 2.7 — Positive values indicate a beneficial effect from Ginkgo
Statistical Analysis 2: Comparison: Ginkgo Exit vs Placebo Exit; Multiple Sclerosis Neuropsychological Questionnaire; Test type: Superiority or Other; p = 0.7, ANCOVA; Mean Difference (Final Values) = 0.8, 95% CI [-3.2 to 4.8], Standard Error of Mean 2 — Positive values indicate a beneficial effect from Ginkgo
Statistical Analysis 3: Comparison: Ginkgo Exit vs Placebo Exit; Community Integration Questionnaire; Test type: Superiority or Other; p = 0.4, ANCOVA; Mean Difference (Final Values) = -0.2, 95% CI [-1.3 to 0.8], Standard Error of Mean 0.6

ADVERSE EVENTS:
Time Frame: Adverse events were collected at 4 weeks, 8 weeks, 12 weeks and 16 weeks (4 weeks after exit).
Description: Subjects reported events. Events were coded according to the Common Terminology Criteria for Adverse Events version 4.
Arm/Group | Placebo | Ginkgo
Serious Adverse Events (participants affected / at risk) | 0/59 | 2/61
Other Adverse Events (participants affected / at risk) | 0/59 | 0/61
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=59) | Ginkgo (N=61)
Myocardial Infarction (Cardiac disorders) | 0 (0) | 1 (1) — Was deemed not related to study intervention
Depression with hospitalization (Psychiatric disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Limitations include underrepresentation of minorities. Subjects overall had mild impairment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes